CLINICAL TRIAL: NCT06802601
Title: The Effect of Visio-Vestibular Exercises Applied in Addition to Manual Therapy and Exercise on Pain, Function, Balance and Reaction Time in Chronic Neck Pain: A Randomized Controlled Study
Brief Title: Effect of Visio-Vestibular Exercises on Pain, Function, Balance, and Reaction Time in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Faruk TANIK, Pt, MSc, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1620
Record Dates: First submitted 2025-01-16; First posted 2025-01-31 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Neck Pain; Chronic Neck Pain
Keywords: Manual Therapy; Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manuel Therapy and Stabilization Exercises (Active Comparator)
  Interventions: Other: Manual Therapy and Exercise
- Manuel Therapy and Stabilization Exercises plus Visio-Vestibular Exercises (Experimental)
  Interventions: Other: Manual Therapy, Exercise and Visio-Vestibular Exercise

INTERVENTIONS:
Other: Manual Therapy and Exercise — Manual Therapy and Exercise
  Arms: Manuel Therapy and Stabilization Exercises
Other: Manual Therapy, Exercise and Visio-Vestibular Exercise — Manual Therapy, Exercise and Visio-Vestibular Exercise
  Arms: Manuel Therapy and Stabilization Exercises plus Visio-Vestibular Exercises

SUMMARY:
The aim of the study was to improve pain, function, balance and reaction times in people with chronic neck pain by stimulating and improving the components that provide input to the central nervous system (proprioceptive, visual, vestibular) through manual therapy and exercise and to reveal the results of vizio-vestibular training applied in addition to manual therapy and exercise. Therefore, the hypotheses of this study were;

H1: Manual therapy and exercise have a positive effect on pain, function, balance and reaction time in people with chronic neck pain.

H2: Vizio-vestibular exercises given in addition to manual therapy and exercise have a positive effect on pain, function, balance and reaction time in people with chronic neck pain.

H3: There is no difference between the effects of manual therapy and exercise and viziovestibular exercises in addition to manual therapy and exercise on pain, function, balance and reaction time in people with chronic neck pain.

DETAILED DESCRIPTION:
Neck pain is defined by the International Association for the Study of Pain (IASP) as pain felt in the area between the occiput and the first thoracic vertebra. Neck pain is a multifactorial disorder and is a major problem in modern society. In 2016, among 154 conditions, low back and neck pain had the highest healthcare expenditure in the United States with an estimated $134.5 billion. In 2012, neck pain was responsible for 25.5 million Americans being absent from work, missing an average of 11.4 days. In 2017, the global age-standardized prevalence and incidence rates of neck pain were 3551.1 and 806.6 per 100,000, respectively.

The cervical spine, especially the upper cervical spine, is the most mobile part of the vertebral column. The highly developed proprioceptive system provides neuromuscular control to the mobile cervical spine and allows efficient utilization of vital organs in the head through unique connections to the vestibular and visual systems. In people with neck pain, disturbances in afferent input from the cervical region may be a possible cause of symptoms such as dizziness, imbalance and visual disturbances, as well as signs of altered postural stability, cervical proprioception and head and eye movement control. For neck pain patients with minimal sensorimotor proprioceptive impairments, conventional treatment approaches may be sufficient. However, clinical experience and research suggest that significant sensorimotor proprioceptive impairments in the cervical spine may be an important factor in the maintenance, relapse or progression of various symptoms in patients with neck pain.

The postural control system includes all sensorimotor and musculoskeletal components involved in the control of 2 important behavioral goals: postural orientation and postural balance. Postural orientation is the relative positioning of body segments relative to each other and to the environment; postural balance is the state in which all forces acting on the body tend to keep the body in a desired position and orientation (static balance) or to move it in a controlled manner (dynamic balance). Postural control provides a stable body platform for efficient execution of goal-directed movements. The somatosensory, vestibular and visual systems are subsystems that provide sensory input to the postural control system.

The Somatosensory System encompasses all mechanoreceptive information from the periphery that leads to the perception of pain, temperature, touch and proprioception. In particular, the proprioceptive system of the cervical spine is highly developed thanks to the large number of mechanoreceptors from the γ-muscle spindles in the deep segmental upper cervical muscles. The γ-muscle spindle system serves as the last common pathway for the regulation of muscle stiffness required for various neuromuscular performances. The dense network of mechanoreceptors in the soft tissues in this region not only controls the movements of each joint, but more importantly, through direct neurophysiological connections to the vestibular and visual systems, informs the Central Nervous System about the orientation of the head relative to the rest of the body. Somatosensory information from the cervical region is the only region with such direct access to the senses of balance and vision.

The Vestibular Subsystem is specifically designed to maintain adequate postural tone in the trunk and limb muscles to ensure overall balance during posture and movement. Neck, eye, trunk and limb muscle reflexes have evolved to meet these requirements. Specialized mechanoreceptors in the semicircular canals become sensitive during changes in the speed of movement, i.e. angular velocity, and specialized mechanoreceptors in the otolith systems of the utricular and saccular maculae provide information about the position and velocity of the head relative to the direction of gravitational forces. Sensory information from the vestibular system is integrated via the vestibular nerve in all the nuclei that make up the vestibular nuclear complex and in the cerebellum.

The Visual Subsystem plays a dominant role in the guidance of movements and this is reflected by the fact that when there is a mismatch between somatosensory inputs and vision, the visual version of events usually prevails. The visual postural system consists of 3 different eye movement systems: the smooth pursuit system, the saccadic system and the optokinetic system. The smooth pursuit system stabilizes images of smoothly moving targets on the fovea with slow eye movements. The saccadic system is responsible for rapid and small movements of both eyes simultaneously when changing a fixation point. The optokinetic system stabilizes images on the entire retina when the entire visual field moves (e.g. when walking).

The aim of the study was to improve pain, function, balance and reaction times in people with chronic neck pain by stimulating and improving the components that provide input to the central nervous system (proprioceptive, visual, vestibular) through manual therapy and exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 18 and 55
2. Complaining of neck pain for at least 3 months or experiencing neck pain at least 2 times in 3 months
3. Volunteering for the study
4. To be able to read and understand Turkish

Exclusion Criteria:

1. Previous history of neck and head trauma or surgery
2. Vertigo or dizziness caused by known or suspected vestibular pathology, ear or brain disorders, sensory nerve pathways (e.g. BPPV) or vascular disorders (e.g. migraine, hypertension)
3. Any musculoskeletal or neurological condition that may affect balance
4. Inflammatory joint disease
5. Cognitive impairment
6. Taking four or more medicines
7. Received physiotherapy treatment for neck pain in the last 12 months
8. People with strabismus, lazy eye and severe refractive errors

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Pain | From enrollment to the end of treatment at week 6. Follow-up assessment 6 weeks after the end of treatment.
  Pain intensity will be questioned with the Visual Analog Scale. The Visual Analog Scale pain assessment scale was first used by Hayes and Patterson in 1921. It measures the severity of pain based on the patient's statement. A straight thin 10 cm line is used. 0 is defined as "no pain" and 10 as "unbearable pain". The patient is asked to mark the point on the line describing the pain. The length of the distance indicates the severity of the patient's pain.
Cervical Range of Motion | From enrollment to the end of treatment at week 6. Follow-up assessment 6 weeks after the end of treatment.
  Goniometric measurement is used in the clinic as an objective measurement tool for the assessment of active range of motion. Goniometer is a durable, simple, easy-to-carry device that can be easily used in almost all joints. Neck flexion, extension, lateral flexion and rotation movements will be evaluated with goniometer.
Function | From enrollment to the end of treatment at week 6. Follow-up assessment 6 weeks after the end of treatment.
  The Neck and Neck Disability Index will be used to assess the level of function in people with neck pain. The questionnaire, whose Turkish validity and reliability study was conducted by Aslan et al. consists of 10 items. Each item is scored from 0 (no disability) to 5 (complete disability). The total score is between 0 (no disability) and 50 (total disability). Disability increases with increasing score and decreases with decreasing score.

SECONDARY OUTCOMES:
Pressure Pain Threshold | From enrollment to the end of treatment at week 6. Follow-up assessment 6 weeks after the end of treatment.
  The pressure value is obtained by pressing a dynamic metal piston with a round disk with a surface area of 1 cm² at its tip into the relevant area. Under the influence of the pressure applied by the metal piston, the hand on the dial moves clockwise. When the algometer leaves the relevant area, the last measured value on the hand is recorded and the zero button is pressed. Thus, the instrument is made ready for further measurements. While applying pressure to the relevant points with the algometer, patients will be asked to say "stop" at the first moment when the feeling of pressure causes discomfort. At the first moment when the patients feel pain, the application of pressure will be stopped and the pressure value at that moment will be recorded. A total of 3 measurements will be made for each marked point with a 30 sec. rest interval between each measurement. Afterwards, the average pressure pain threshold values will be recorded. In this direction, the Trapezius, Biceps Brachi
Balance | From enrollment to the end of treatment at week 6. Follow-up assessment 6 weeks after the end of treatment.
  Static, eyes open-eyes closed and stability limits will be evaluated with a computerized balance device. The device consists of a computer and a balance platform. The individual will be asked to step on the platform barefoot and step on the designated areas. For static balance with eyes open and eyes closed, the individual will be asked to stand on the device for 30 seconds without speaking and moving as stably as possible. Balance results with eyes open and eyes closed will be recorded in square millimeters and anteroposterior and medio-lateral deviation values will be recorded in millimeters. For the stability limit, it will be asked to try to reach 4 different points by transferring the body weight in 4 different directions in a 360-degree circle on the screen. The limits he/she can reach will be recorded in degrees.
Reaction Time | From enrollment to the end of treatment at week 6. Follow-up assessment 6 weeks after the end of treatment.
  Reaction time measurements of the upper extremities will be performed on the dominant side, non-dominant side and bilaterally with the "Test You Brain Pro" system. Measurements will be made with the help of a device containing visual/auditory and perceptual/cognitive tasks. Using a program with sound, light and variable timer, the participant will be asked to follow the stimuli, hand contact with the light will be monitored and the time until the program ends will be recorded.
The Cervical Flexor Endurance Test | From enrollment to the end of treatment at week 6. Follow-up assessment 6 weeks after the end of treatment.
  The Cervical Flexor Endurance Test is a test that measures the endurance of participants' deep neck flexors. The participant lies supine on the bed without a pillow. The participant is asked to keep the occiput 2.5 cm above the bed while maintaining the neck position. When the participant starts the test, the time is started and stopped when the participant cannot control the occiput.
Cervical Extensor Endurance Test | From enrollment to the end of treatment at week 6. Follow-up assessment 6 weeks after the end of treatment.
  The cervical extensor endurance test aims to be able to determine the weakness of both the superficial and deep neck extensors. With the participant lying prone, the head and neck past the edge of the table and the cervicothoracic region stabilized, the patient is asked to maintain a neutral head position. At the beginning of the test, the test is timed with a chronimeter and terminated when the participant is unable to maintain the position.
Quality of Life | From enrollment to the end of treatment at week 6. Follow-up assessment 6 weeks after the end of treatment.
  The Short Form-36 (SF-36) is a test consisting of 8 sub-parameters and 36 items that the participant fills in and answers by himself/herself to obtain information about the health status of the person. Scoring is based on 100 points and the scores are between 0 and 100 points for each sub-parameter. "0" is calculated as the worst value and '100' as the best value.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi Univeristy, Izmir, Cigli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guitton D, Kearney RE, Wereley N, Peterson BW. Visual, vestibular and voluntary contributions to human head stabilization. Exp Brain Res. 1986;64(1):59-69. doi: 10.1007/BF00238201. PMID 3490396
- [Background] Kristjansson E, Treleaven J. Sensorimotor function and dizziness in neck pain: implications for assessment and management. J Orthop Sports Phys Ther. 2009 May;39(5):364-77. doi: 10.2519/jospt.2009.2834. PMID 19411769